CLINICAL TRIAL: NCT02973035
Title: Effect of Add-on of Amlodipine Versus Valsartan on Diastolic Dysfunction Associated With Hypertension
Brief Title: Amlodipine Versus Valsartan for Improvement of Diastolic Dysfunction Associated With Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Yuhan Corporation (Industry)
Responsible Party: Principal Investigator, Duk-Hyun Kang, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YMC016
Record Dates: First submitted 2016-11-22; First posted 2016-11-25 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Amlodipine; Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amlodipine (Experimental): Amlodipine 2.5mg added to antihypertensive therapy
  Interventions: Drug: Amlodipine
- Valsartan (Experimental): Valsartan 40mg added to antihypertensive therapy
  Interventions: Drug: Valsartan

INTERVENTIONS:
Drug: Amlodipine
  Arms: Amlodipine
Drug: Valsartan
  Arms: Valsartan

SUMMARY:
Hypertensive patients are at increased risk of developing LV hypertrophy and myocardial fibrosis, which cause diastolic dysfunction. Because the activation of rennin-angiotensin-aldosterone system (RAAS) has been shown to induce LV hypertrophy and myocardial fibrosis, the RAAS may play a central role in the pathogenic process from hypertension to diastolic HF. Inhibitors of RAAS have been considered as a treatment option for these patients, and the angiotensin receptor blockers (ARB) have been of interest because they antagonize the effects of angiotensin II more completely. However, the Irbesartan in Heart Failure with Preserved Systolic Function (I-PRESERVE) trial reported that treatment with irbesartan did not reduce the risk of death or hospitalization for cardiovascular causes among 4,128 patients who had HF with a preserved LV ejection fraction. The degree of improvement of diastolic dysfunction was associated with the extent of systolic blood pressure reduction, whether a RAAS inhibitor or non-RAAS blood pressure lowering was used. Amlodipine is a potent and well-tolerated calcium channel blocker, and seems to be appropriate for achieving more aggressive systolic blood pressure target and improving diastolic dysfunction in hypertensive patients, because amlodipine is clinically very useful for controlling systolic blood pressure. Assessment of diastolic function by echocardiography will be helpful to determine whether addition of amlodipine or an ARB to standard therapy is more beneficial to hypertensive patients with diastolic dysfunction. The investigators hypothesize that amlodipine added to standard therapy will be superior to valsartan in improving diastolic dysfunction by lowering systolic blood pressure more effectively in hypertensive patients, and try to examine this hypothesis in a prospective, open-label, randomized comparison study using blinded echocardiographic evaluation for end point.

DETAILED DESCRIPTION:
Approximately half of hypertensive patients have diastolic dysfunction and diastolic dysfunction is associated with development of congestive heart failure and increased mortality. The Framingham study reported that 51% of patients with HF have a preserved left ventricular (LV) ejection fraction and hypertension is the strongest risk factor for HF with preserved ejection fraction, also termed diastolic heart failure. The rates of death and morbidity in these patients are as high as in patients with HF and a low LV ejection fraction. Hypertensive patients are at increased risk of developing LV hypertrophy and myocardial fibrosis, which cause relaxation abnormality and decreased compliance of LV with a rise in the LV diastolic pressure. Although diastolic HF associated with hypertension is a clinically significant problem, few clinical trials have been conducted and there is no proven pharmacological therapy to improve outcomes. Because the activation of rennin-angiotensin-aldosterone system (RAAS) has been shown to induce LV hypertrophy and myocardial fibrosis, the RAAS may play a central role in the pathogenic process from hypertension to diastolic HF. Inhibitors of RAAS have been considered as a treatment option for these patients, and the angiotensin receptor blockers (ARB) have been of interest because they antagonize the effects of angiotensin II more completely. However, the Irbesartan in Heart Failure with Preserved Systolic Function (I-PRESERVE) trial reported that treatment with irbesartan did not reduce the risk of death or hospitalization for cardiovascular causes among 4,128 patients who had HF with a preserved LV ejection fraction.

The degree of improvement of diastolic dysfunction was associated with the extent of systolic blood pressure reduction, whether a RAAS inhibitor or non-RAAS blood pressure lowering was used. The Systolic Blood Pressure Intervention Trial (SPRINT) compared the benefit of treatment of systolic blood pressure to a target of less than 120 mmHg with treatment to a target of less than 140 mmHg, and recently reported that targeting a systolic blood pressure of less than 120 mmHg, as compared with less than 140 mmHg, resulted in lower rates of fatal and nonfatal major cardiovascular events and all-cause death. Amlodipine is a potent and well-tolerated calcium channel blocker, and seems to be appropriate for achieving more aggressive systolic blood pressure target and improving diastolic dysfunction in hypertensive patients, because amlodipine is clinically very useful for controlling systolic blood pressure. Evaluating the effect of treatments on diastolic dysfunction has been limited by difficulties in non-invasive measure of LV diastolic pressure, but recent advances in echocardiography have made it possible to assess diastolic dysfunction accurately and reproducibly. Thus, assessment of diastolic function by echocardiography will be helpful to determine whether addition of amlodipine or an ARB to standard therapy is more beneficial to hypertensive patients with diastolic dysfunction. To the best of our knowledge, there has been no randomized trial to compare the effect of amlodipine versus an ARB on improving diastolic dysfunction in hypertensive patients. The investigators hypothesize that amlodipine added to standard therapy will be superior to valsartan in improving diastolic dysfunction by lowering systolic blood pressure more effectively in hypertensive patients, and try to examine this hypothesis in a prospective, open-label, randomized comparison study using blinded echocardiographic evaluation for end point.

ELIGIBILITY:
Inclusion Criteria:

* Controlled hypertension: systolic BP < 150 and diastolic BP < 90 mmHg in persons aged 60 years or older, systolic BP < 140 and diastolic BP < 90 mmHg in persons 40 through 59 years according to the JNC 8th guideline
* Evidence of diastolic dysfunction showing E/E' > 10
* The patient agrees to the study protocol and the schedule of clinical and echocardiographic follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site

Exclusion Criteria:

* Unwillingness or inability to comply with the procedures described in this protocol
* Planned cardiac surgery or planned major non-cardiac surgery within the study period.
* Stroke or coronary revascularization in the past 6 months.
* Clinically significant pulmonary disease.
* Untreated hyperthyroidism, or hypothyroidism.
* A diagnosis of cancer (other than superficial squamous or basal cell skin cancer) in the past 3 years or current treatment for the active cancer.
* Female of child-bearing potential who do not use adequate contraception and women who are pregnant or breast-feeding
* Any clinically significant abnormality identified at the screening visit, physical examination, laboratory tests, or electrocardiogram which, in the judgment of the Investigator, would preclude safe completion of the study.
* LV ejection fraction < 50%.
* Significant renal disease manifested by serum creatinine > 2.5 mg/dL
* Hepatic disease or biliary tract obstruction, or significant hepatic enzyme elevation (ALT or AST > 3 times upper limit of normal).
* History of intolerance to ARB or amlodipine.
* Hypertrophic or restrictive cardiomyopathy.
* Moderate or severe valvular disease.
* Constrictive pericarditis
* Atrial fibrillation with a heart rate > 120/min.
* Sitting systolic BP < 100 mmHg

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2016-12; Primary Completion 2020-01-06 (Actual); Study Completion 2020-01-06 (Actual)

PRIMARY OUTCOMES:
Change in the ratio of E velocity (Early mitral inflow velocity) to E' velocity (Early mitral annular velocity) | 24 weeks

SECONDARY OUTCOMES:
Change in systolic blood pressure | 24 weeks
Change in global LV longitudinal strain | 24 weeks
Change in LV mass | 24 weeks
Change in left atrial volume | 24 weeks
Change in clinical composite | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Duk-Hyun Kang, M.D., Principal Investigator — Asan Medical Center
Locations (4):
- South Korea (4):
  - Busan Baik Hospital, Busan
  - Busan University Hospital, Busan
  - Chungnam University Hospital, Daejeon
  - Asan Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No